CLINICAL TRIAL: NCT01830764
Title: An Open-label Safety and Tolerability Study of LTS 0.3% With Red Light Applied to the Backs of Healthy Volunteers
Brief Title: Open-label Safety and Tolerability Study of LTS-PDT in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS-ACN06
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Red light dose (PDT) 75 J/cm2 (Other): Subjects in Cohort 1 will receive active and vehicle solution followed by a red light dose of 75 J/cm2 at 25 mW/cm2
  Interventions: Drug: Red Light (PDT)
- Red Light (PDT) 150 J/cm2 (Other): Subjects in Cohort 2 will receive active and vehicle solution followed by a red light dose of 150 J/cm2 at 40 mW/cm2
  Interventions: Drug: Red Light (PDT)

INTERVENTIONS:
Drug: Red Light (PDT) — LTS, 0.3% applied topically followed by red light dose (75 J/cm2 or 150 J/cm2)
  Other Names: LTS-PDT

SUMMARY:
The purpose of this study is assess the safety and tolerability of lemuteporfin topical solution (LTS) with exposure to red light (PDT), when applied to the backs of healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label, safety study in healthy volunteers. Two cohorts, of 6 subjects each, will be enrolled (total subjects = 12). Each subject will have test areas identified on the back and receive a single LTS, vehicle solution and red light (PDT) applied to the test areas on the back. Subjects will be followed for safety at study visits occurring on Day 1 (baseline and treatment), Day 2, and Day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 18 years of age or older
2. Fitzpatrick skin types I-IV

Exclusion Criteria:

1. Current pregnancy or lactation.
2. Presence of severe facial acne, acne fulminans or conglobata, or nodulocystic acne.
3. Poor skin condition on the back, including erythema, dryness, sunburn, dermatological malignancies, infections, cuts, abrasions, tattoo, excess of hair or any other skin condition
4. Subjects who have used any agents known to produce significant photosensitivity reactions (tetracyclines, phenothiazines, trimethoprim, etc.) within 2 weeks of Day 1 or 5 half-lives, whichever is longer.
5. Subjects who have used any medicated topical therapy on the back within 3 days of Day 1.
6. Chronic treatment with low dose aspirin, a non-steroidal anti inflammatory drug (NSAID), or an anticoagulant regimen such as warfarin (Coumadin).
7. Abnormal findings on screening ECG deemed clinically significant by the Investigator.
8. Active participation in an experimental therapy study or experimental therapy within 30 days of Day 1.
9. Screening clinical chemistry or hematology laboratory value that is considered clinically significant, in the opinion of the Investigator.
10. Subjects who are a poor medical risk because of other systemic diseases or active uncontrolled infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 1 week
  Adverse events and local tolerability assessed at pre and immediately post treatment, at Day 1 and Day 7 following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Dosik, MD, Principal Investigator — TKL Research Inc (Research Clinics Division)
Locations (1):
- TKL Research Inc (Research Clinics Division), Paramus, New Jersey, United States